CLINICAL TRIAL: NCT01628562
Title: A Comparison of the Perioperative Hemodynamic Effects of Remifentanil and Esmolol: a Double Blind Randomized Controlled Study
Brief Title: A Comparison of the Perioperative Hemodynamic Effects of Remifentanil and Esmolol in Intracranial Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dilek Esmolol
Record Dates: First submitted 2012-05-28; First posted 2012-06-27 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2012-12

CONDITIONS: Tachycardia; Hypertension; Myocardial Ischemia
Keywords: Remifentanil; Esmolol; Intracranial surgery; Heart rate; Blood pressure
MeSH Terms: conditions — Tachycardia; Hypertension; Myocardial Ischemia | interventions — esmolol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GroupE/Esmolol infusion (Active Comparator): Heart rate control, Beta blocker
  Interventions: Drug: Esmolol
- GroupR/Remifentanil infusion (Experimental): Heart rate control, opioid
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Esmolol — Esmolol 50 mcg/kg/min
  Other Names: Brevibloc
  Arms: GroupE/Esmolol infusion
Drug: Remifentanil — Remifentanil 0.5 mcg/kg/min
  Other Names: Ultiva
  Arms: GroupR/Remifentanil infusion

SUMMARY:
It was hypothesized that the use of esmolol as an alternative to remifentanil with sevoflurane inhalation anesthesia during intracranial surgery, could provide better hemodynamic conditions and cause lesser side effects in the perioperative period. It was the main objective of this study to compare the effect of esmolol and remifentanil on the incidence of tachycardia and hypertension and the intraoperative fentanyl consumption. The comparison of postoperative troponine I and creatine phosphokinase levels and EKG changes were the secondary objectives.

DETAILED DESCRIPTION:
During neurosurgical procedures intubation, insertion of the head pins, extubation and the early postoperative period are the time lines in which cerebral autoregulation can be impaired by changes in heart rate and blood pressure. Several anesthetic regimens have been implied to overcome this problem. Remifentanil is used in neurosurgery since it allows early recovery and neurologic evaluation. Esmolol on the other hand is also very short acting, effective to blunt cardiovascular responses during surgery and has no significant effect on intracranial pressure and cerebral blood flow. In addition esmolol is addressed to reduce perioperative ischemia during noncardiac surgery.

It was hypothesized that the use of esmolol as an alternative to remifentanil with sevoflurane inhalation anesthesia during intracranial surgery, could provide better hemodynamic conditions and cause lesser side effects in the perioperative period. It was the main objective of this study to compare the effect of esmolol and remifentanil on the incidence of tachycardia and hypertension and the intraoperative fentanyl consumption. The comparison of postoperative troponine I and creatine phosphokinase levels and EKG changes were the secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial surgery

Exclusion Criteria:

* heart rate ≤ 50,
* atrioventricular block,
* sick sinus syndrome,
* heart failure,
* history of asthma,
* hypertension,
* impaired renal or hepatic function,
* patients receiving beta blockers or calcium channel blockers,
* emergency surgery.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
It is the main objective of this study to compare the effect of esmolol and remifentanil on the incidence of tachycardia and hypertension | during intubation, head pin insertion, extubation, early postoperative period

SECONDARY OUTCOMES:
the intraoperative fentanyl consumption | during intubation, head pin insertion, extubation, early postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazicioglu, Principal Investigator — MD
Locations (2):
- Turkey (Türkiye) (2):
  - Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey
  - Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara

REFERENCES:
- [Background] Heinke W, Zysset S, Hund-Georgiadis M, Olthoff D, von Cramon DY. The effect of esmolol on cerebral blood flow, cerebral vasoreactivity, and cognitive performance: a functional magnetic resonance imaging study. Anesthesiology. 2005 Jan;102(1):41-50. doi: 10.1097/00000542-200501000-00010. PMID 15618785
- [Background] Landoni G, Turi S, Biondi-Zoccai G, Bignami E, Testa V, Belloni I, Cornero G, Zangrillo A. Esmolol reduces perioperative ischemia in noncardiac surgery: a meta-analysis of randomized controlled studies. J Cardiothorac Vasc Anesth. 2010 Apr;24(2):219-29. doi: 10.1053/j.jvca.2009.07.008. Epub 2009 Oct 2. PMID 19800816